CLINICAL TRIAL: NCT03786315
Title: Exploring 'VOLITION' in Context - a Study to Inform the Implementation of a New Intervention
Acronym: VOLITION
Status: Completed | Type: Observational
Sponsor: University of Exeter (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University of Leeds (Other)
Responsible Party: Sponsor
Other Study IDs: 1819/06; 253014 (Other: IRAS)
Record Dates: First submitted 2018-11-22; First posted 2018-12-26 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Decision Making; Aged; Multimorbidity; General Practice
Keywords: Primary care; Elderly; Older age; Multimorbidity; Shared decision-making; Patient involvement
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Usual care: Older patients with multimorbidity and the GPs with whom they consult, from across five GP practices in Devon

SUMMARY:
Trial Design

A mixed-methods sequential explanatory approach in general practices, using quantitative questionnaire data followed by qualitative interviews.

Trial Participants

Patients aged 65 years and above with more than one long-term health problem (multimorbidity); and the GPs that these patients consult with.

Planned Sample Size

5 GP practices; 15 GPs; 150 patients

Planned study period:

01/01/21 - 30/12/21; 1 year

Objectives

Primary

To establish the determinants of adoption, implementation and maintenance of the critical, core components of the VOLITION intervention, designed to be embedded within GP consultations, and to determine those components of VOLITION that can be tailored to ensure that the intervention is modifiable in context.

Secondary

To describe the current context of GP consultations for older patients with multimorbidity in England, including current innovations, in light of recent organisational changes as a result of the COVID-19 pandemic.

To describe the effect of recent changes to the context of GP consultations (towards remote consulting) on patients' and GPs' perceptions of shared decision-making To investigate factors which could potentially influence the successful implementation of interventions such as VOLITION in the context of remote vs. face-to-face consultations.

The Intervention 'VOLITION':

* half-day training workshop for GPs in shared decision-making
* written involvement-facilitating tool for patients (delivered by post and available in the waiting room).

DETAILED DESCRIPTION:
1 BACKGROUND

The VOLITION intervention was developed to facilitate the involvement of older people with multimorbidity in clinical decision-making during general practice consultations.The overarching project follows the Intervention Mapping framework as a means of systematically applying existing literature and relevant theory to each step of intervention development and evaluation.

There are two core intervention components:

* A patient tool, in the form of a leaflet, to facilitate patients to convey their preferences for involvement to the GP
* A workshop for GPs, to train them in shared decision-making orientated communication skills, delivered in the context of the challenges facing GPs when consulting with this patient group

To enable transparency and sustainability in complex intervention development it is important to theorise the context in which intervention mechanisms will work. Further research is required to determine the factors affecting the incorporation of patients' priorities and preferences during clinical decision-making in the context of remote GP consultations for older people with multimorbidity. This study will inform the final iteration of 'VOLITION' ahead of testing the intervention in a randomised controlled pilot study.

3 OBJECTIVES AND OUTCOME MEASURES/ENDPOINTS

The aim of this study is:

To establish the determinants for future adoption, implementation and maintenance of the VOLITION intervention, and to determine those components of VOLITION that can be tailored to ensure that the intervention is modifiable in context.

To describe the current modalities of GP consultations for older patients with multimorbidity in England, including any existing innovations to improve quality and access to GP consultations for this patient group, in light of recent organisational changes as a result of the COVID-19 pandemic.

To describe the effect of recent changes to the modality of GP consultations (towards remote consulting) on patients' and GPs' perceptions of shared decision-making.

To investigate factors which could potentially influence the future implementation and evaluation of VOLITION in the context of remote vs. face-to-face consultations.

4 STUDY DESIGN

A mixed methods sequential explanatory study undertaken in UK general practices. Quantitative questionnaire data will be collected first. Qualitative interview data will then be used to explain, build, and elaborate on the quantitative findings by exploring participants' views in more depth. Questionnaire data will inform the purposive selection of patient participants. The quantitative and qualitative phases are therefore connected in the intermediate stage of the study, prior to the interpretation of the combined findings.

5 STUDY SETTING

Five GP practices will be recruited from Devon, UK. Recruitment of local practices will be prioritised in order to reduce travel expenses for the research team and with the aim of shortening the recruitment period. However, to obtain sociodemographic diversity in the participant sample, practices will be recruited from both rural and urban areas.

A minimum practice size of 3,000 patients will ensure sufficient numbers of eligible participants. (It is anticipated that there will be approximately 800 older patients with multimorbidity in an average 8,000 patient practice.

7 STUDY PROCEDURES

7.1 Sampling

An average of three (total = 15 GPs), and at least 2, GPs per practice will be recruited. Patients aged 65 and above with known multimorbidity, defined as the presence of two or more long-term conditions, will be approached.

Patient participants will be identified using an automated practice database search strategy designed by the research team. Recruited GPs will use this 'flag' to identify ten consecutive potential participants from their working schedule. Random sampling of patients is not required as the clinical presentations, and therefore the nature of the decision-making between consecutive consultations, is expected to be random. A total of 150 (minimum 100) potential patients will be identified across five practices, with the aim of obtaining data from at least half of these patients.

The sample size is sufficient to allow for the estimation of standard deviations for the clinical outcome measures being tested and to tentatively report between-group differences in outcomes by mode of consultation (e.g. face-to-face vs. remote). It is also sufficient to obtain a purposively selected sub-sample of participants for qualitative interviews.

7.2 Recruitment

Drop-out and loss to follow-up will be taken into account at patient, GP or practice level by over-recruiting. Practices will receive an email followed by telephone correspondence inviting their participation. Practice recruitment will be dependent on an expression of interest from at least two of their GPs. Practices will be incentivised through payment for local coordination, set-up, and for GPs' time and workload. Payments were determined by advisors from the South West Clinical Research Network.

For each recruited GP, ten potential patient participants with consecutive GP contacts, for any mode of consultation (telephone, video, eConsult or face-to-face), will be screened by GPs using pre-specified eligibility criteria (see eligibility form) at the time of consultation. Eligibility data will be collected anonymously. If eligible, GPs will label patient packs to be sent by post following the consultation. Eligible patients will receive a cover letter, participant information sheet* and a post-consultation questionnaire with a pre-paid envelope for return to the research team. Using the questionnaire, patients will indicate their consent to be contacted for a subsequent telephone interview with the researcher and they will be asked to provide their contact information. Patients who do not wish to participate will not be expected to return their questionnaire. All recruited GPs will also be asked to complete a post-consultation questionnaire and to participate in a telephone interview.

7.3 Consent

Written consent from GPs will be obtained at the time of practice recruitment. Consent to identify and approach potential patient participants will be obtained from the practice manager. Consent from patients, to use their questionnaire data, will be confirmed by return of questionnaires and patients will be advised of this using the Participant Information Sheet. Written consent will be obtained prior to telephone interviews, informed by an interim telephone call to clarify procedures and to answer participant's questions, by return of consent forms in pre-paid envelopes. Verbal consent will also be confirmed before commencing interviews. If stated, reasons for declining to participate in interviews will be recorded anonymously. Identifiable data will not be accessed without prior patient consent.

7.4 Baseline data

Practice level data (list size, location and deprivation, practice size, staffing, rural/urban) and GP participant data (age, gender, ethnicity and time since qualification) will be collected at the time of recruitment. Information will be requested from practices regarding whether, and how, they have identified, or addressed, the potential for inequality in experience of remote consultations for the patient group of interest.

Data will be obtained at practice level regarding the mode (phone, video, eConsult or face-to-face) and relative frequency of consultations with older patients with multimorbidity. A template will be provided to GP surgeries in order to collect and compare data regarding each practice's interpretation and delivery of remote vs. face-to-face consulting and how GPs' workload is being managed in respect of these. Data will be obtained from GPs, at the time of recruitment, regarding their preferences for the different consultation modalities when consulting with older patients with multimorbidity.

Patient demographics (age, gender and ethnicity) and health status data will be collected via self-report using post-consultation questionnaires. An electronic frailty index score, for each patient where applicable, will be obtained from GPs on post-consultation questionnaires.

7.5 Study assessments

Quantitative outcome measure data

The General Practice Patient Survey (GPPS) uses five-point Likert scales. A subset of these are appropriate for evaluation of Patient Reported Outcome Measures (PROMs) on the post-consultation patient questionnaires. PROMs will be used to collect data on patients' preferences for involvement in decision-making, the extent to which patients felt engaged in decision-making, the patient's preferred mode of consultation and whether they obtained this, their satisfaction with the care received, whether they felt they were given enough time, and a measure of patient enablement.

A post-consultation questionnaire for GPs will collect data regarding the mode and approximate duration (using a scale) of consultation and GPs' ratings of the extent to which they felt they involved the patient in decision-making.

Qualitative interview data

Following receipt and initial analysis of post-consultation participant questionnaires, twenty patients will be sampled and twice this number will be approached. Patients will be selected purposively and iteratively, using questionnaire data to ensure heterogeneity by age, sociodemographic characteristics and health status, and also by mode of consultation received, preferences for and experiences of shared decision-making. Patients will be contacted by telephone to arrange an interview. All participating GPs (n = 10-15) will be invited by email. The sample size will be reviewed when assessing thematic saturation.

Semi-structured telephone interviews will be aided by a topic guide and will be digitally audio recorded, transcribed and supported by field notes. Following initial open discussion, the topic guide will encourage participants to discuss the reasoning behind their questionnaire responses. For example, participants may be prompted to discuss their ratings of shared decision-making, or their preferences for a particular consultation modality, in greater depth. The intervention will be described to participants (see topic guide in Appendix) at a suitable mid-point during telephone interviews, in order to stimulate discussion regarding factors that could potentially affect the implementation of VOLITION. Participants will be prompted to discuss these factors in the context of different consultation modalities and in light of ongoing social distancing measures in the UK. Intervention materials will not be posted to patients in advance of interviews so as to avoid the influence of materials on the earlier interview dialogue. Participants will be encouraged to discuss their own ideas in order to collect fresh data without the influence of the researcher. Audio recordings of participant interviews will be coded using Nvivo computer software.

Mixed methods

Data analysis will take a sequential-explanatory approach .The quantitative questionnaire data and subsequent analysis (see details below) will provide a general understanding of participants' perspectives on the research problem. The qualitative data and their analysis will refine and explain the statistical results by exploring purposively selected participants' views in more depth. Interpretation of interviews will combine both deductive and inductive methods to investigate whether the theory developed earlier in the project holds, but also being open to new data and emerging themes. The concept of thematic saturation will be applied and negative cases will be actively sought. The consistency with which the coding is applied will be assessed on a fifth of the data.

ELIGIBILITY:
Inclusion criteria:

* GP practice located in Devon, UK
* GP participants must be permanent practice employees
* Patient participants must be aged 65 and above with multimorbidity

Exclusion criteria:

* Previous participation in the focus group study to refine the intervention
* Locum GPs
* Trainee GPs and junior doctors working in general practice
* Temporarily registered patients
* Vulnerable patients (as screened by usual GP)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older patients (aged 65 and above) and the GPs that they consult with
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
Factors potentially influencing the future successful implementation and evaluation of VOLITION | 2 months
  Questionnaire & interviews with data integration Qualitative data
  Common themes from the analysis of interview data regarding the perceived impact of the changes towards remote consulting, on patients and on GPs, will be reported. Significant divergent themes will be actively sought.
  Data integration
  Interview findings will be presented in line with the purposive sampling (informed by participant questionnaire data). Findings may therefore be interpreted in the context of participant characteristics, or by consultation modality, for example. Where interview themes provide greater depth regarding findings from questionnaire items, the interpretation of these findings will be discussed in the context of existing literature and previously developed theory. Reporting will be designed with a view to informing future policy and interventions to support older people with multimorbidity during remote consultations.

SECONDARY OUTCOMES:
The current context of GP consultations for older patients with multimorbidity | 2 months
  Descriptive & qualitative data
The effect of recent changes to the context of GP consultations on perceptions of shared decision-making | 2 months
  Questionnaire & interviews with data integration

CONTACTS AND LOCATIONS:
Overall Officials: Jo Butterworth, MRCGP, Principal Investigator — University of Exeter Medical School
Locations (1):
- University of Exeter Medical School, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abraham, C. (2012) Designing and evaluating interventions to change health-related behaviour patterns. In I. Boultron and P.M.D. Ravaud (Eds.), Randomized Clinical Trials of Nonpharmacological Treatments. (pp. 357-368). London: Chapman and Hall.
- [Background] Arain M, Campbell MJ, Cooper CL, Lancaster GA. What is a pilot or feasibility study? A review of current practice and editorial policy. BMC Med Res Methodol. 2010 Jul 16;10:67. doi: 10.1186/1471-2288-10-67. PMID 20637084
- [Background] Barnett K, Mercer SW, Norbury M, Watt G, Wyke S, Guthrie B. Epidemiology of multimorbidity and implications for health care, research, and medical education: a cross-sectional study. Lancet. 2012 Jul 7;380(9836):37-43. doi: 10.1016/S0140-6736(12)60240-2. Epub 2012 May 10. PMID 22579043
- [Background] Barr PJ, Thompson R, Walsh T, Grande SW, Ozanne EM, Elwyn G. The psychometric properties of CollaboRATE: a fast and frugal patient-reported measure of the shared decision-making process. J Med Internet Res. 2014 Jan 3;16(1):e2. doi: 10.2196/jmir.3085. PMID 24389354
- [Background] Bartholomew, L.K., Parcel, G.S., Kok, G., Gottlieb, N.H., Fernandez, M.E. (2011) Planning health promotion programs: an intervention mapping approach. London: Willey Press.
- [Background] Berkelmans PG, Berendsen AJ, Verhaak PF, van der Meer K. Characteristics of general practice care: what do senior citizens value? A qualitative study. BMC Geriatr. 2010 Nov 2;10:80. doi: 10.1186/1471-2318-10-80. PMID 21044316
- [Background] Berwick DM, Nolan TW, Whittington J. The triple aim: care, health, and cost. Health Aff (Millwood). 2008 May-Jun;27(3):759-69. doi: 10.1377/hlthaff.27.3.759. PMID 18474969
- [Background] Bowling A, Rowe G, McKee M. Patients' experiences of their healthcare in relation to their expectations and satisfaction: a population survey. J R Soc Med. 2013 Apr;106(4):143-9. doi: 10.1258/jrsm.2012.120147. PMID 23564898
- [Background] Bowling A. An "inverse satisfaction law"? Why don't older patients criticise health services? J Epidemiol Community Health. 2002 Jul;56(7):482. doi: 10.1136/jech.56.7.482-a. No abstract available. PMID 12080150
- [Background] Bunn F, Goodman C, Manthorpe J, Durand MA, Hodkinson I, Rait G, Millac P, Davies SL, Russell B, Wilson P. Supporting shared decision-making for older people with multiple health and social care needs: a protocol for a realist synthesis to inform integrated care models. BMJ Open. 2017 Feb 7;7(2):e014026. doi: 10.1136/bmjopen-2016-014026. PMID 28174225
- [Background] Burt J. Following the mixed methods trail: some travel advice. Br J Gen Pract. 2015 May;65(634):264-5. doi: 10.3399/bjgp15X685045. No abstract available. PMID 25918329
- [Background] Butterworth JE, Campbell JL. Older patients and their GPs: shared decision making in enhancing trust. Br J Gen Pract. 2014 Nov;64(628):e709-18. doi: 10.3399/bjgp14X682297. PMID 25348995
- [Background] Campbell J, Hobbs FD, Irish B, Nicholson S, Pringle M, Reeve J, Rosenthal J. UK academic general practice and primary care. BMJ. 2015 Jul 31;351:h4164. doi: 10.1136/bmj.h4164. No abstract available. PMID 26231511
- [Background] Campbell JL, Fletcher E, Britten N, Green C, Holt TA, Lattimer V, Richards DA, Richards SH, Salisbury C, Calitri R, Bowyer V, Chaplin K, Kandiyali R, Murdoch J, Roscoe J, Varley A, Warren FC, Taylor RS. Telephone triage for management of same-day consultation requests in general practice (the ESTEEM trial): a cluster-randomised controlled trial and cost-consequence analysis. Lancet. 2014 Nov 22;384(9957):1859-1868. doi: 10.1016/S0140-6736(14)61058-8. Epub 2014 Aug 3. PMID 25098487
- [Background] Campbell J, Smith P, Nissen S, Bower P, Elliott M, Roland M. The GP Patient Survey for use in primary care in the National Health Service in the UK--development and psychometric characteristics. BMC Fam Pract. 2009 Aug 22;10:57. doi: 10.1186/1471-2296-10-57. PMID 19698140
- [Background] Coleman T. Using video-recorded consultations for research in primary care: advantages and limitations. Fam Pract. 2000 Oct;17(5):422-7. doi: 10.1093/fampra/17.5.422. PMID 11021903
- [Background] Couet N, Desroches S, Robitaille H, Vaillancourt H, Leblanc A, Turcotte S, Elwyn G, Legare F. Assessments of the extent to which health-care providers involve patients in decision making: a systematic review of studies using the OPTION instrument. Health Expect. 2015 Aug;18(4):542-61. doi: 10.1111/hex.12054. Epub 2013 Mar 4. PMID 23451939
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Croker JE, Swancutt DR, Roberts MJ, Abel GA, Roland M, Campbell JL. Factors affecting patients' trust and confidence in GPs: evidence from the English national GP patient survey. BMJ Open. 2013 May 28;3(5):e002762. doi: 10.1136/bmjopen-2013-002762. PMID 23793686
- [Background] Croker J.E. and Campbell J.L. (2009) 'Satisfaction with access to healthcare: qualitative study of rural patients and practitioners' Primary Healthcare Research & Development, vol. 10, pp. 309-319.
- [Background] Department of Health (2013) Liberating the NHS: No decision about me, without me, [Online], Available: https://www.gov.uk/government/uploads/system/uploads/attachment_data/file/216980/Liberating-the-NHS-No-decision-about-me-without-me-Government-response.pdf [02 Nov 2015].
- [Background] Department of Health (2012) Long Term Conditions Compendium of Information: Third Edition, [Online], Available: https://www.gov.uk/government/uploads/system/uploads/attachment_data/file/216528/dh_134486.pdf [02Nov 2015].
- [Background] Department of Health (2011) Atlas of variation, [Online], Available: https://www.rightcare.nhs.uk/index.php/atlas/atlas-of-variation-2011 [02 Nov 2015].
- [Background] Department of Health (2001) National Service Framework for Older People, [Online], Available: https://www.gov.uk/government/publications/quality-standards-for-care-services-for-older-people [02 Nov 2015].
- [Background] Drennan V, Walters K, Lenihan P, Cohen S, Myerson S, Iliffe S; SPICE Research Group. Priorities in identifying unmet need in older people attending general practice: a nominal group technique study. Fam Pract. 2007 Oct;24(5):454-60. doi: 10.1093/fampra/cmm034. Epub 2007 Aug 4. PMID 17675658
- [Background] Eldridge, S. and Kerry, S. (2012) A Practical Guide to Cluster Randomised Trials in Health Services Research, 1st Edition, New Jersey USA: Wiley.
- [Background] Elwyn G, Hutchings H, Edwards A, Rapport F, Wensing M, Cheung WY, Grol R. The OPTION scale: measuring the extent that clinicians involve patients in decision-making tasks. Health Expect. 2005 Mar;8(1):34-42. doi: 10.1111/j.1369-7625.2004.00311.x. PMID 15713169
- [Background] Elwyn G, Edwards A, Kinnersley P, Grol R. Shared decision making and the concept of equipoise: the competences of involving patients in healthcare choices. Br J Gen Pract. 2000 Nov;50(460):892-9. PMID 11141876
- [Background] Fisher JD, Fisher WA. Changing AIDS-risk behavior. Psychol Bull. 1992 May;111(3):455-74. doi: 10.1037/0033-2909.111.3.455. PMID 1594721
- [Background] Flocke SA, Miller WL, Crabtree BF. Relationships between physician practice style, patient satisfaction, and attributes of primary care. J Fam Pract. 2002 Oct;51(10):835-40. PMID 12401151
- [Background] Friedman R, Sobel D, Myers P, Caudill M, Benson H. Behavioral medicine, clinical health psychology, and cost offset. Health Psychol. 1995 Nov;14(6):509-18. doi: 10.1037//0278-6133.14.6.509. PMID 8565925
- [Background] Glaser, B.G. and Strauss, A.L. (1967) The discovery of grounded theory, Chicago, IL: Aldine.
- [Background] Green, J. and Thorogood, N. (2009) Qualitative methods for health research, 2nd Edition, California USA: Sage.
- [Background] Hardeman W, Sutton S, Griffin S, Johnston M, White A, Wareham NJ, Kinmonth AL. A causal modelling approach to the development of theory-based behaviour change programmes for trial evaluation. Health Educ Res. 2005 Dec;20(6):676-87. doi: 10.1093/her/cyh022. Epub 2005 Mar 21. PMID 15781446
- [Background] Herbert RD, Bo K. Analysis of quality of interventions in systematic reviews. BMJ. 2005 Sep 3;331(7515):507-9. doi: 10.1136/bmj.331.7515.507. PMID 16141160
- [Background] Noel PH, Parchman ML, Williams JW Jr, Cornell JE, Shuko L, Zeber JE, Kazis LE, Lee AF, Pugh JA. The challenges of multimorbidity from the patient perspective. J Gen Intern Med. 2007 Dec;22 Suppl 3(Suppl 3):419-24. doi: 10.1007/s11606-007-0308-z. PMID 18026811
- [Background] Homa L, Rose J, Hovmand PS, Cherng ST, Riolo RL, Kraus A, Biswas A, Burgess K, Aungst H, Stange KC, Brown K, Brooks-Terry M, Dec E, Jackson B, Gilliam J, Kikano GE, Reichsman A, Schaadt D, Hilfer J, Ticknor C, Tyler CV, Van der Meulen A, Ways H, Weinberger RF, Williams C. A participatory model of the paradox of primary care. Ann Fam Med. 2015 Sep;13(5):456-65. doi: 10.1370/afm.1841. PMID 26371267
- [Background] Iliffe S, Lenihan P, Orrell M, Walters K, Drennan V, Tai SS; SPICE Research Team. The development of a short instrument to identify common unmet needs in older people in general practice. Br J Gen Pract. 2004 Dec;54(509):914-8. PMID 15588536
- [Background] Johnson BT, Scott-Sheldon LA, Carey MP. Meta-synthesis of health behavior change meta-analyses. Am J Public Health. 2010 Nov;100(11):2193-8. doi: 10.2105/AJPH.2008.155200. Epub 2010 Feb 18. PMID 20167901
- [Background] Kiesler DJ, Auerbach SM. Optimal matches of patient preferences for information, decision-making and interpersonal behavior: evidence, models and interventions. Patient Educ Couns. 2006 Jun;61(3):319-41. doi: 10.1016/j.pec.2005.08.002. Epub 2005 Dec 20. PMID 16368220
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Background] Legare F, Stacey D, Turcotte S, Cossi MJ, Kryworuchko J, Graham ID, Lyddiatt A, Politi MC, Thomson R, Elwyn G, Donner-Banzhoff N. Interventions for improving the adoption of shared decision making by healthcare professionals. Cochrane Database Syst Rev. 2014 Sep 15;(9):CD006732. doi: 10.1002/14651858.CD006732.pub3. PMID 25222632
- [Background] Levinson W, Kao A, Kuby A, Thisted RA. Not all patients want to participate in decision making. A national study of public preferences. J Gen Intern Med. 2005 Jun;20(6):531-5. doi: 10.1111/j.1525-1497.2005.04101.x. PMID 15987329
- [Background] Loh A, Leonhart R, Wills CE, Simon D, Harter M. The impact of patient participation on adherence and clinical outcome in primary care of depression. Patient Educ Couns. 2007 Jan;65(1):69-78. doi: 10.1016/j.pec.2006.05.007. PMID 17141112
- [Background] Marengoni A, Angleman S, Melis R, Mangialasche F, Karp A, Garmen A, Meinow B, Fratiglioni L. Aging with multimorbidity: a systematic review of the literature. Ageing Res Rev. 2011 Sep;10(4):430-9. doi: 10.1016/j.arr.2011.03.003. Epub 2011 Mar 23. PMID 21402176
- [Background] May CR, Mair F, Finch T, MacFarlane A, Dowrick C, Treweek S, Rapley T, Ballini L, Ong BN, Rogers A, Murray E, Elwyn G, Legare F, Gunn J, Montori VM. Development of a theory of implementation and integration: Normalization Process Theory. Implement Sci. 2009 May 21;4:29. doi: 10.1186/1748-5908-4-29. PMID 19460163
- [Background] McCabe R, John P, Dooley J, Healey P, Cushing A, Kingdon D, Bremner S, Priebe S. Training to enhance psychiatrist communication with patients with psychosis (TEMPO): cluster randomised controlled trial. Br J Psychiatry. 2016 Dec;209(6):517-524. doi: 10.1192/bjp.bp.115.179499. Epub 2016 Jul 21. PMID 27445354
- [Background] McCabe, R., et al. (2015). Shared Decision Making in Dementia: The ShareD Project, [online], Available: http://medicine.exeter.ac.uk/research/healthserv/shared/ [14 Nov 2015].
- [Background] McAllister M, Dunn G, Payne K, Davies L, Todd C. Patient empowerment: the need to consider it as a measurable patient-reported outcome for chronic conditions. BMC Health Serv Res. 2012 Jun 13;12:157. doi: 10.1186/1472-6963-12-157. PMID 22694747
- [Background] McBride D, Hardoon S, Walters K, Gilmour S, Raine R. Explaining variation in referral from primary to secondary care: cohort study. BMJ. 2010 Nov 30;341:c6267. doi: 10.1136/bmj.c6267. PMID 21118873
- [Background] McHugh ML. Interrater reliability: the kappa statistic. Biochem Med (Zagreb). 2012;22(3):276-82. PMID 23092060
- [Background] Melzer D, Tavakoly B, Winder RE, Masoli JA, Henley WE, Ble A, Richards SH. Much more medicine for the oldest old: trends in UK electronic clinical records. Age Ageing. 2015 Jan;44(1):46-53. doi: 10.1093/ageing/afu113. Epub 2014 Aug 7. PMID 25103030
- [Background] Michie, S., Johnston, M., Francis, J., Hardeman, W., Eccles, M. (2008) 'From theory to intervention: mapping theoretically derived behavioural determinants to behaviour change techniques', Applied Psychology, vol. 57, no. 4, Oct, pp. 660-680.
- [Background] Michie S, Johnston M, Abraham C, Lawton R, Parker D, Walker A; "Psychological Theory" Group. Making psychological theory useful for implementing evidence based practice: a consensus approach. Qual Saf Health Care. 2005 Feb;14(1):26-33. doi: 10.1136/qshc.2004.011155. PMID 15692000
- [Background] Moher D, Schulz KF, Altman DG. The CONSORT statement: revised recommendations for improving the quality of reports of parallel-group randomised trials. Lancet. 2001 Apr 14;357(9263):1191-4. PMID 11323066
- [Background] Moore GF, Audrey S, Barker M, Bond L, Bonell C, Hardeman W, Moore L, O'Cathain A, Tinati T, Wight D, Baird J. Process evaluation of complex interventions: Medical Research Council guidance. BMJ. 2015 Mar 19;350:h1258. doi: 10.1136/bmj.h1258. PMID 25791983
- [Background] Mujica-Mota RE, Roberts M, Abel G, Elliott M, Lyratzopoulos G, Roland M, Campbell J. Common patterns of morbidity and multi-morbidity and their impact on health-related quality of life: evidence from a national survey. Qual Life Res. 2015 Apr;24(4):909-18. doi: 10.1007/s11136-014-0820-7. Epub 2014 Oct 26. PMID 25344816
- [Background] NHS Information Centre. (2009) Trends in consultation rates in general practice 1995 to 2008: analysis of the Q Research® database [online], Available: https://catalogue.ic.nhs.uk/publications/primary-care/general-practice/tren-cons-rate-gene- prac-95-09/tren-cons-rate-gene-prac-95-09-95-08-rep.pdf [03 Nov 2015].
- [Background] Oeppen J, Vaupel JW. Demography. Broken limits to life expectancy. Science. 2002 May 10;296(5570):1029-31. doi: 10.1126/science.1069675. No abstract available. PMID 12004104
- [Background] Ommen O, Thuem S, Pfaff H, Janssen C. The relationship between social support, shared decision-making and patient's trust in doctors: a cross-sectional survey of 2,197 inpatients using the Cologne Patient Questionnaire. Int J Public Health. 2011 Jun;56(3):319-27. doi: 10.1007/s00038-010-0212-x. Epub 2010 Nov 13. PMID 21076932
- [Background] Pawson, R. and Tilley, M. (1997) Realistic Evaluation, London: Sage.
- [Background] Peters RM. Matching physician practice style to patient informational issues and decision-making preferences. An approach to patient autonomy and medical paternalism issues in clinical practice. Arch Fam Med. 1994 Sep;3(9):760-3; discussion 764. doi: 10.1001/archfami.3.9.760. PMID 7987509
- [Background] Petticrew M. Why certain systematic reviews reach uncertain conclusions. BMJ. 2003 Apr 5;326(7392):756-8. doi: 10.1136/bmj.326.7392.756. No abstract available. PMID 12676848
- [Background] Price EL, Bereknyei S, Kuby A, Levinson W, Braddock CH 3rd. New elements for informed decision making: a qualitative study of older adults' views. Patient Educ Couns. 2012 Mar;86(3):335-41. doi: 10.1016/j.pec.2011.06.006. Epub 2011 Jul 14. PMID 21757315
- [Background] Richards, D.A. and Hallberg, I.R. (2015) Complex Interventions in Health. An overview of research methods. 1st edition, Abingdon UK: Routledge.
- [Background] Royal College of General Practitioners (2013). The 2022 GP Compendium of Evidence, [online], Available: http://www.rcgp.org.uk/~/media/Files/Policy/A-Z-policy/The-2022-GP-Compendium-of-Evidence.ashx [20 Oct 2015].
- [Background] Saba GW, Wong ST, Schillinger D, Fernandez A, Somkin CP, Wilson CC, Grumbach K. Shared decision making and the experience of partnership in primary care. Ann Fam Med. 2006 Jan-Feb;4(1):54-62. doi: 10.1370/afm.393. PMID 16449397
- [Background] Salisbury C, Johnson L, Purdy S, Valderas JM, Montgomery AA. Epidemiology and impact of multimorbidity in primary care: a retrospective cohort study. Br J Gen Pract. 2011 Jan;61(582):e12-21. doi: 10.3399/bjgp11X548929. PMID 21401985
- [Background] Steel N, Hardcastle AC, Clark A, Mounce LT, Bachmann MO, Richards SH, Henley WE, Campbell JL, Melzer D. Self-reported quality of care for older adults from 2004 to 2011: a cohort study. Age Ageing. 2014 Sep;43(5):716-20. doi: 10.1093/ageing/afu091. Epub 2014 Jul 11. PMID 25015897
- [Background] Tarrant C, Stokes T, Baker R. Factors associated with patients' trust in their general practitioner: a cross-sectional survey. Br J Gen Pract. 2003 Oct;53(495):798-800. PMID 14601357
- [Background] Tate AR, Nicholson A, Cassell JA. Are GPs under-investigating older patients presenting with symptoms of ovarian cancer? Observational study using General Practice Research Database. Br J Cancer. 2010 Mar 16;102(6):947-51. doi: 10.1038/sj.bjc.6605593. Epub 2010 Mar 2. PMID 20197770
- [Background] Taylor AH, Thompson TP, Greaves CJ, Taylor RS, Green C, Warren FC, Kandiyali R, Aveyard P, Ayres R, Byng R, Campbell JL, Ussher MH, Michie S, West R. A pilot randomised trial to assess the methods and procedures for evaluating the clinical effectiveness and cost-effectiveness of Exercise Assisted Reduction then Stop (EARS) among disadvantaged smokers. Health Technol Assess. 2014 Jan;18(4):1-324. doi: 10.3310/hta18040. PMID 24433837
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] The Cochrane Collaboration. (2011) Cochrane Handbook of Systematic Reviews, [online], Available: http://handbook.cochrane.org/ [03 Nov 2015].
- [Background] The Equator Network (2015). Enhancing the QUAlity and Transparency Of health Research, [online], Available: http://www.equator-network.org/ [27-10-2015].
- [Background] Tong A, Sainsbury P, Craig J. Consolidated criteria for reporting qualitative research (COREQ): a 32-item checklist for interviews and focus groups. Int J Qual Health Care. 2007 Dec;19(6):349-57. doi: 10.1093/intqhc/mzm042. Epub 2007 Sep 14. PMID 17872937
- [Background] van den Brink-Muinen A, van Dulmen SM, de Haes HC, Visser AP, Schellevis FG, Bensing JM. Has patients' involvement in the decision-making process changed over time? Health Expect. 2006 Dec;9(4):333-42. doi: 10.1111/j.1369-7625.2006.00413.x. PMID 17083560
- [Background] Wetzels R, Harmsen M, Van Weel C, Grol R, Wensing M. Interventions for improving older patients' involvement in primary care episodes. Cochrane Database Syst Rev. 2007 Jan 24;2007(1):CD004273. doi: 10.1002/14651858.CD004273.pub2. PMID 17253501
- [Background] WILLIAMSON J, STOKOE IH, GRAY S, FISHER M, SMITH A, MCGHEE A, STEPHENSON E. OLD PEOPLE AT HOME. THEIR UNREPORTED NEEDS. Lancet. 1964 May 23;1(7343):1117-20. doi: 10.1016/s0140-6736(64)91803-3. No abstract available. PMID 14132624
- [Background] Wong, G., Westhorp, R., Pawson, R., Greenhalgh, T. (2013) Realist synthesis RAMESES training materials, [online], Available: http://www.ramesesproject.org/media/Realist_reviews_training_materials.pdf [24 Oct 2015].
- [Background] World Health Organization (2016). Definition of an older or elderly person, [online}, Available: http://www.who.int/healthinfo/survey/ageingdefnolder/en/ [13/10/2016]
- [Background] World Health Organization (1994). A declaration on the promotion of patients' rights in Europe, [online], Available: http://www.who.int/genomics/public/eu_declaration1994.pdf [03 Nov 2015].
- [Derived] Butterworth J, Richards S, Warren F, Pitchforth E, Campbell J. Randomised feasibility trial and embedded qualitative process evaluation of a new intervention to facilitate the involvement of older patients with multimorbidity in decision-making about their healthcare during general practice consultations: the VOLITION study protocol. Pilot Feasibility Stud. 2020 Oct 26;6:161. doi: 10.1186/s40814-020-00699-7. eCollection 2020. PMID 33117558